CLINICAL TRIAL: NCT05251597
Title: Comparison of the Effects of Green Exercise Programs Including Resistance Exercises and Aerobic Exercises on Metabolic Syndrome Parameters in Elderly Individuals
Brief Title: Comparison of the Effects of Green Exercise Programs on Metabolic Syndrome Parameters in Elderly Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Green exercise
Record Dates: First submitted 2021-12-23; First posted 2022-02-22 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; exercise; geriatrics
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized
Who Masked: Participant
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- green exercise group-1 (aerobic) (Experimental): Forty participants who meet the inclusion criteria will first be given warm-up exercises for 10 minutes, then walking at a moderate intensity (65% of heart rate) for 40 minutes and then stretching exercises for 5 minutes
  Interventions: Other: green exercise with aerobic exercise
- green exercise group-2 (aerobic+resistance) (Experimental): For 40 participants who met the inclusion criteria, first 10 minutes of warm-up exercises, then 20 minutes of moderate-intensity (65% of heart rate) walking, followed by 10 minutes of low-intensity (50% of the maximum repetitions) and 10 minutes of high-intensity (80% of the maximum repetitions) resistance exercises will be applied in the presence of a physiotherapist. resistance exercises; shoulder flexors and abductors, elbow flexors and extensors, hip flexors and extensors, knee flexors and extensors, hip abductor muscle group will be performed. At the end of each session, 5 minutes of stretching exercises will also be applied.
  Interventions: Other: green exercise with aerobic exercise
- Control group (No Intervention): The exercise program will not be implemented. Evaluations will be made at the beginning and end of the study.

INTERVENTIONS:
Other: green exercise with aerobic exercise — Green exercise is a type of exercise done outdoors. It is an advantageous type of exercise in benefiting from sunlight and reducing anxiety. It is mostly applied in the form of brisk walking in the open air.
  Other Names: green exercise with aerobic and resistance exercises
  Arms: green exercise group-1 (aerobic); green exercise group-2 (aerobic+resistance)

SUMMARY:
The aim of this study is to compare the effects of exercise programs that only aerobic exercise and combination aerobic exercise and resistance exercises on the metabolic syndrome parameters in the green exercise concept.

DETAILED DESCRIPTION:
One hundred twenty volunteer participants aged 65 years over will be included in the study. Participants will be randomly divided into three groups as aerobic, aerobic and resistance and control group. While a group will receive only aerobic exercise, the other group group will receive both aerobic and resistance exercises and one of the group will receive no exercise. Exercises will be held in an open and green area. At the beginning of the treatment and at the end of the twelfth week Hemoglobin A1c (HbA1c), Triglyceride, Hdl cholesterol, Ldl cholesterol, total cholesterol and blood glucose will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* people aged over 65 years
* Be fit to participate in exercise program after the first cardiac examination by the physician
* Individuals whose blood lipids, Hg a1c and glucose values were checked within 3 months
* According to the International Physical Activity Assessment Questionnaire, those who are physically inactive
* Having a score above 24 in the Minimental Test

Exclusion Criteria:

* Having neuromuscular disease
* Serious medical condition (for example, advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.)
* Having an orthopedic disease that interferes with walking
* Having a score below 24 in the Minimental Test

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-10-08 (Estimated); Study Completion 2022-11-12 (Estimated)

PRIMARY OUTCOMES:
physical activity level | Change from baseline physical activity level at week 12.
  physical activity level will be evaulated with international physical activity questionnairre (IPAQ). The questionnaire is based on calculating the MET (metabolic equivalent) value spent by evaluating at least 10 minutes of physical activity in the last seven days in terms of frequency, duration (minutes) and intensity. According to this questionnaire, physical activity level is categorized into 4 classes: inactive, not active enough, active, very active.
blood pressure | Change from baseline blood pressure at week 12.
  Systolic and diastolic blood pressure will be measured using a standard semi-automatic sphygmomanometer.
hemoglobin A1c | Change from baseline hemoglobin A1c at week 12.
  After 12-14 hr of fasting, a 10 cc blood sample will be collected from each participant. HbA1c will be measured using the Chromatography method with a com-mercial kit .
lipid profile | Change from baseline lipid profile at week 12.
  HDL cholesterol, LDL cholesterol, total cholesterol and triglyceride serum levels will be measured to evaluate the lipid profile.HDL cholesterol, LDL cholesterol, total cholesterol and triglyceride will be assessed using enzymatic colorimetry with commercial kits.
fasting blood glucose | Change from baseline fasting blood glucose at week 12.
  After 12-14 hr of fasting, a 10 cc blood sample will be collected from each participant. Fasting blood samples from the antecubital vein will be collected by vacuum tubes. For biochemical analysis, Fasting blood glucose will be assessed with a commercial kit.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University, Istanbul
  - Emel Mete, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayaz EY, Dincer B, Cinbaz G, Karacan E, Benli RK, Mete E, Bilgic H, Mesci B. The Effect of Exercise on Spexin and Follistatin in Elderly Individuals. J Cachexia Sarcopenia Muscle. 2025 Feb;16(1):e13692. doi: 10.1002/jcsm.13692. PMID 39895162